CLINICAL TRIAL: NCT05336825
Title: The Application of External Fractional CO2 Laser Energy Versus Topical Lidocaine for the Treatment of Vestibulodynia in Premenopausal Women on Hormonal Contraception: a Pilot Study
Brief Title: CO2 Laser vs Lidocaine for Vestibulodynia in Premenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlantic Health System (Other)
Collaborators: Foundation for Morristown Medical Center (Unknown)
Responsible Party: Principal Investigator, Michael Ingber, Director of The Center for Specialized Women's Health, division of Garden State Urology/Atlantic Health System, Atlantic Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GSU-MLT001
Record Dates: First submitted 2022-04-13; First posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Vulvodynia
MeSH Terms: conditions — Vulvodynia | interventions — Lasers, Gas

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- CO2 laser (Experimental): Mona Lisa CO2 laser will be applied externally to the vulvar vestibule in three sessions over a three month period.
  Interventions: Device: CO2 laser
- Lidocaine (Active Comparator): 5% topical lidocaine will be applied nightly via a cotton square in participants
  Interventions: Drug: Lidocaine patch 5%

INTERVENTIONS:
Device: CO2 laser — Mona Lisa CO2 laser
  Arms: CO2 laser
Drug: Lidocaine patch 5% — lidocaine
  Arms: Lidocaine

SUMMARY:
CO2 laser energy is currently used widely for the treatment of postmenopausal women who have vaginal atrophy due to the lack of estrogen. However, its effect on premenopausal women with hormonally-mediated vulvar vestibulodynia is unknown. This study seeks to evaluate the effect of CO2 laser on young women and compare it to topical lidocaine.

DETAILED DESCRIPTION:
The purpose of this study is to see if vaginal laser therapy with MonaLisa Touch® will be more effective in treating vestibulodynia than current treatment with a topical lidocaine ointment. Vestibulodynia is a common bothersome condition and is more likely to occur in women on hormonal contraceptive treatment. To date, there are no effective treatments that address the underlying causes of the disease. MonaLisa Touch® is a laser procedure that delivers CO2 laser energy to the vaginal wall tissue. This energy causes the patient's own body to regenerate collagen and blood vessels, changing the tissue to make it healthier. The MonaLisa Touch® technology may help vestibulodynia by potentially fixing the underlying cause. This may be more effective than using the topical lidocaine which makes the tissue numb.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years to 40 years
* Hormonal contraceptive therapy for at least one year consecutive duration
* Vestibulodynia diagnosis meeting the following criteria:

  * Localized vulvar pain to vaginal vestibule
  * At least 3 months duration
  * Without clear identifiable cause

Exclusion Criteria:

* Suspected primary cause to vestibular pain that warrants directed treatment
* History of chronic infection or autoimmune disease
* Prior pelvic surgery including mesh placement for incontinence or prolapse, vestibulectomy, vulvectomy, or labiaplasty
* Active vulvar or vaginal infection
* Allergy or contraindication to topical lidocaine treatment
* Prior diagnosis or treatment of vulvar intraepithelial neoplasia or vulvar malignancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
VAS | 3 months
  visual analog pain scale to q-tip palpation

SECONDARY OUTCOMES:
PFDI | 3 months
  pelvic floor distress inventory

CONTACTS AND LOCATIONS:
Locations (1):
- Garden State Urology, Denville, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No